CLINICAL TRIAL: NCT06211465
Title: Cardiovascular And Metabolic Risk After Arthroplasty: the CAMERA Study
Brief Title: Cardiovascular And Metabolic Risk After Arthroplasty
Acronym: CAMERA
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Collaborators: Tartu University Hospital (Other); Estonian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Kaspar Tootsi, Orthopedic research fellow, University of Tartu
Other Study IDs: 296T-14
Record Dates: First submitted 2020-12-30; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee; Osteoarthritis of the Hip; Cardiovascular Diseases; Metabolic Syndrome
Keywords: metabolomics; arthroplasty; cardiovascular risk; arterial stiffness
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Cardiovascular Diseases; Metabolic Syndrome | interventions — Arthroplasty, Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with end-stage osteoarthritis (OA), who were eligible for total joint arthroplasty in Tartu University Hospital. Exclusion criteria: posttraumatic OA, infectious or endocrine arthropathy, acute or chronic inflammatory disease, malignancies, end-stage renal impairment (eGFR < 60ml/min/1.73m2), dysrhythmias, clinically relevant heart failure, heart valve-disease, diabetes.
  Interventions: Procedure: Total joint arthroplasty
- Controls: Gender and age matched control group, who is recruited from the general practitioner (GP) list and who are from the same geographical regions as the cases. Excluding criteria: acute or chronic inflammatory disease, GP visitation due to hip or knee problems, persistent knee or hip pain, diabetes, symptomatic coronary disease, dysrhythmias, cerebrovascular or peripheral artery disease, malignancy or renal impairment.

INTERVENTIONS:
Procedure: Total joint arthroplasty — Hip or knee total joint arthroplasty
  Groups: Cases

SUMMARY:
Osteoarthritis is a chronic joint disease that lacks curative therapy. Epidemiological studies show increase in the burden of disease. Total joint arthroplasty is one of the best treatment options for end-stage osteoarthritis. However, the specific effects of total joint arthroplasty on cardiovascular risk and metabolic profile are largely unknown. The aim of this project is to elucidate how hip and knee total joint arthroplasty impacts cardiovascular risk and metabolomic profile in comparison with general population. We hypothesize that arthroplasty decreases pain, systemic inflammation levels and increases functional status that all lead to decreased metabolic and cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria for the arthroplasty group:

primary hip and knee OA (according to the American College of Rheumatology criteria) eligible for total joint arthroplasty

Exclusion Criteria for the arthroplasty group:

posttraumatic OA, infectious and endocrine related arthropathy, any acute or chronic inflammatory disease, malignancy, renal insufficiency (estimated glomerular filtration rate (eGFR) < 60ml/min/1.73m2), cardiac arrhythmia, clinically significant heart failure, valvular disease, diabetes.

Exclusion criteria for the control group:

any concomitant acute or chronic inflammatory disease, a visit to family practitioner due to hip or knee joint complaints, any persistent knee or hip joint pain, diabetes, symptomatic coronary artery disease, cardiac arrhythmia, cerebrovascular or peripheral artery disease, malignancies and renal insufficiency.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Aortic pulse wave velocity at 5 years after arthroplasty | 5 years
  5 years after the beginning of study for control group; measurements are done using the Sphygmocor device.

SECONDARY OUTCOMES:
Changes in low-molecular weight metabolites | 5 years
  Low-molecular weight metabolites are measured using Biocrates Absolute IDQ p180 kit (BIOCRATES Life Sciences AG, Innsbruck, Austria), which enables to quantify lipides, acylcarnitines, aminoacids, biogenic amines, polyamides
Oxidative stress index | 5 years
  Serum oxidative stress index. Expressed in %. The percentage of the ratio of total plasma peroxide concentration to plasma total antioxidative capacity (TAC, expressed in mmol trolox equivalent/L).
Leptin levels | 5 years
  Measured from serum. Expressed in ng/ml.
Metabolic syndrome risk score | 5 years
  A composite risk score is used to assess metabolic syndrome risk and include waist circumference(cm), HDL-cholesterol level(mmol/L), fasting glucose level(mmol/L), triglycerides level(mmol/L), blood pressure(mmHg). Each factor gives one point to the total score (range 0-5)
Harris Hip score or Hospital for Special Surgery Knee score | 5 years
  Harris Hip Score for hip arthroplasty patients. The HHS is divided into three sections. The first section are questions about pain and its impact which are answered by the patient or client. The second and third sections require specialist to assess the patient or client's hip joint and function. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Central systolic blood pressure | 5 years
  Central systolic blood pressure is measured using the Sphygmocor device. Expressed in mmHg.
Central diastolic blood pressure | 5 years
  Central diastolic blood pressure is measured using the Sphygmocor device. Expressed in mmHg.
Composite of cardiovascular clinical events | 5 years
  Composite of stroke, myocardial infarction, cardiovascular death, unstable angina
Oxidized LDL-cholesterol | 5 years
  Measured from serum. Expressed in mmol/L
Adiponectin level | 5 years
  Measured from serum, expressed in ng/ml
Augmentation index | 5 years
  Measured using the Sphygmocor device. The augmentation index (AI) is an indirect measure of arterial stiffness and increases with age, and it is calculated as AG (augmentation pressure) divided by PP(pulse pressure) ×100 to give a percentage.
SF-36 | 5 years
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Hospital for Special Surgery knee score | 5 years
  The HSS Knee Score is based on a total of 100 points. The score is divided into seven categories, which include pain, function, range of motion, muscle strength, flexion deformity, instability, and subtractions. The knee is initially given a score of 0, and additions or subtractions are made according to specific criteria. The higher the score, the better the outcome. Approximately 50% of the score is based on a patient interview and the remaining on physical exam.
Central pulse pressure | 5 years
  Measured using the Sphygmocor device. Expressed in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Kaspar Tootsi, PhD, MD, Principal Investigator — University of Tartu; Kadri Vilba, MD, Study Chair — University of Tartu; Aare Märtson, PhD, MD, Study Chair — University of Tartu; Jaak Kals, PhD, MD, Study Chair — University of Tartu
Locations (1):
- University of Tartu, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No